CLINICAL TRIAL: NCT02501941
Title: Spreading Depolarization and Ketamine Suppression
Acronym: SAKS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Andrew Phillip Carlson, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15-056
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cortical Spreading Depolarization; Cortical Spreading Depression; Subarachoid Hemorrhage; Traumatic Brain Injury
Keywords: Ketamine; Cortical Spreading Depolarization; Cortical Spreading Depression
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine first (Experimental): Randomization to receive ketamine as first post-operative sedative in the Neuroscience Intensive Care unit. This group will cross-over to "other sedation" after 6 hours, then alternate every 6 hours between these groups during the entirety of invasive neuromonitoring.
  Interventions: Drug: ketamine
- Other sedation (typically propofol) first (Experimental): Randomization to receive sedative other than ketamine as first post-operative sedative in the Neuroscience Intensive Care unit. This group will cross-over to ketamine after 6 hours, then alternate every 6 hours between these groups during the entirety of invasive neuromonitoring.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — Ketamine will be used as a sedative alternative to other more conventional sedatives (such as propofol, versed, or dexmedetomidine) in 6 hour blocks of time. Ketamine will be titrated at the bedside based on clinically desired Riker Sedation-Agitation Scale target. Both groups will receive the drug in this multiple crossover design. The only difference between groups is which sedation regimen is started first to minimize any bias related to differences in physiology in the early post-operative phase.

SUMMARY:
Hypothesis: Cortical spreading depolarizations are inhibited by the NMDA receptor antagonist Ketamine Aim 1: To demonstrate, in a group of patients with acute severe brain injury requiring surgery including traumatic brain injury and aneurysmal subarachnoid hemorrhage, whether use of continuous infusion of ketamine decreases frequency of occurrence of cortical spreading depolarizations.

DETAILED DESCRIPTION:
Cortical spreading depolarizations (CSD) are massive events which recently have been observed in many types of acute brain injury and likely lead to expansion of injury. These "brain tsunamis" are unlike any other type of brain electrical event (such as seizures or normal neuronal transmission) in that they progress very slowly across the surface of the brain (2-5mm/minute) and involve near complete depolarization of the neurons and other cells. The only similar event in neurophysiology is an anoxic depolarization, which is the final wave of loss of cell function preceding death in cells suffering severe, irreversible hypoxia or ischemia(1). In the case of CSD, the cell is able to recover function, however, at an enormous metabolic expense. Massive amounts of energy substrate (ATP, glucose, oxygen) as well as the delivery system to bring these substrates (blood flow) are required to restore the normal ionic gradient of the cell membrane and cell function. Because of this loss of function of cells, normal electrocortical (ECog) activity is transiently lost, resulting in a depression of the high frequency cortical activity, which is why the phenomenon is also frequently referred to as "cortical spreading depression." CSD has been definitively documented to occur after many types of acute brain injury including ischemic stroke, aneurysmal subarachnoid hemorrhage, intracerebral hemorrhage, and severe traumatic brain injury(2,3). The true incidence is, for the time being, unknown, in that the measurement technique requires placement of a small cortical electrode at the time of a surgical procedure. This limits the region of measurement to relatively small area in patients undergoing surgery, however even in this very small sample, the incidence of delayed SD after brain injury ranges from 53-88%(4). Efforts are underway to attempt to measure CSD less invasively(5) or non-invasively(6,7), however these techniques are currently under exploration and do not have the robust reliability of the cortical electrode system.

Mounting human data coupled with extensive animal data supports the assertion that CSD is not only a marker in response to severe brain injury, but in fact, plays a causal role in injury propagation(8). Animal data is fairly definitive in this assertion, in that CSD can be studied in uninjured brain and inducing CSD leads to neuronal death, particularly with repeated events. Note the progressive loss of brain electrical activity with repeated CSD in the figure to the right. In animal models, CSD clearly leads to expansion of injury, particularly in ischemic stroke models. Human data is unavoidably observational to this point, however by observing multiple physiologic modalities, the deleterious effects become clear. A spectrum of local blood flow responses to CSD have been observed, ranging from a wave of hyperemia (termed the normal hemodynamic response) to a wave of ischemia (termed the inverse hemodynamic response(9, 10)). The factors that determine the response likely have to do with the availability of substrate (glucose, oxygen) and delivery (blood flow) coupled with the baseline metabolic state of the tissue (depressed metabolic state may be more resistant). When the inverse hemodynamic response is observed, an associated wave of tissue hypoxia is observed, which becomes linearly more hypoxic with repeated CSD in a short interval(11). Brain metabolism also can be measured during CSD, and consistent metabolic challenge is noted, with increased micro dialysis lactate and decreased glucose(12). In the case of repeated events, this glucose depletion becomes progressive due to inadequate time for the tissue to recover between these massive events leading to progressive ischemia(12).

From a clinical perspective, the metabolic data can support a deleterious effect, but the effect on clinical outcome is critical in determining if the events are relevant as a potential target for therapy. The occurrence and severity of CSD has been closely linked to both development of new stroke as well as clinical outcome in both retrospective and prospective series. In subarachnoid hemorrhage, Dreier(13) reported a direct association with clinical delayed ischemic neurologic defect (DIND) and the presence of a cluster of SD. Furthermore, in this small series, the patients who went on to develop stroke had markedly longer periods of depression, indicating inability of the tissue to recover from the event compared to patients without delayed stroke. The most extensive clinical outcome data is from traumatic brain injury (TBI)(14,15) where the presence of any CSD showed a non-significant trend toward predicting worse outcome, however CSD occurring in already dysfunctional tissue (termed isoelectric spreading depolarization or ISD) was stronger predictor of clinical outcome than a composite score of most standard variables through to predict outcome (OR 7.58 (95%CI 2.64-21.8) for ISD compared to 1.76(95%CI 1.26-2.46) for the composite prognostic score)(15).

This mounting observational data as to the deleterious effects of CSD has led to increased excitement regarding CSD as a novel target for prevention of delayed injury after diverse types of acute brain injury(16). The optimal target or agent has not been defined, but there are promising animal data supporting a wide variety of agents, primarily targeting NMDAVR, as this is thought to be an important factor in propagation of SD(17). Initial clinical case reports of the effect of ketamine being used as sedation in patients with severe TBI(18) led to a larger scale effort to retrospectively study the various anesthetics used for standard clinical care on the frequency of CSD in monitored patients(19). Using only the sedation medications for which there were >1000 cumulative hours of ECog recording while on that medication, the effects of propofol, fentanyl, midazolam, ketamine, morphine, and sufentanyl were examined. The study found a consistent effect of ketamine in decreased probability of CSD/h per patient. This was nearly linearly dose dependent, and importantly, in multivariate analysis, ketamine still emerged as having a significant effect on decreasing both occurrence of CSD as well as the occurrence of the more deleterious clusters of CSD(19).

Though ongoing observational data is still clearly needed to better characterize the susceptibility and effects of CSD, in order to move toward trial of CSD directed therapy, a prospective trial of the effect of ketamine on the occurrence of CSD is necessary to confirm these retrospective observations and establish the precedent for future therapeutic trials. The SAKS trial will provide important confirmatory pilot data to direct the implementation of future trials.

This is a prospective, randomized, controlled, multiple cross-over trial evaluating the efficacy of ketamine in the suppression of CSDs. This multiple crossover design was chosen in order to be able to develop preliminary data which could guide implementation of future multicenter trials. Because of the significant variability between patients, a study randomized by patients would be subject to a large amount of potential bias. Because factors such as time of day or hospital day also are known to affect CSD, a brief crossover period of 6 hours was chosen. The study will be registered with clinicaltrials.gov prior to enrollment of patients. Patients with severe traumatic brain injury or subarachnoid hemorrhage who fit the inclusion/exclusion criteria will be approached by either research coordinators or study investigators who will consent the LAR for the study prior to clinically indicated craniotomy. It is not expected that patients will be able to independently consent given the severity of the condition, however, if the patient is conscious, attempts will be made to discuss the study with him or her as well.

The patient's surgical procedure will be carried out as planned. The only alteration of the surgical procedure will be the placement of a subdural electrode strip (1x6 cortical strip: Integra: Plainsboro, NJ) on the brain cortex adjacent to the operative site at the end of the procedure. These strips are standard, FDA approved, disposable, pre-sterilized devices used routinely for epilepsy monitoring. In addition, the investigators have used these strips as part of our post-injury IRB approved protocol (10-159) for many days after surgery. The cortical strip (plus a dermal reference electrode on the mastoid or apex of the skull) will be monitored with a Moberg CNS monitor. (Moberg Research, Ampler, PA).The Moberg monitor is a modified version of a standard clinical use multiparametric monitoring system shown below which was cleared by the FDA in 2008. The only difference is the ECog amplifier, which allows for direct full frequency spectrum DC recording.

Upon arrival, post-operatively, to the Neurosciences Intensive Care Unit, the patient will have randomization completed via online randomization program. Randomization will be to allocate patients to either of two groups: 1) Ketamine first or 2) Propofol/other first. No secondary randomization criteria are thought to be necessary given the small sample size for this pilot trial. Initiation of the protocoled sedation regimen will begin on the next hour divisible by 6 (i.e. 06:00, 12:00, 18:00, 24:00). The randomization will determine which sedative to start, and after that the ketamine and propofol/other infusions will be alternated every 6 hours on the above schedules.

Dosages of these sedating medications will not be standardized, but rather titrated to clinical effect. The clinical effect will be determined by the attending intensivist based on the patient's clinical needs. This level of sedation will be communicated to nursing via the Riker Sedation-Agitation Score(20). A minimal dose of ketamine (0.1mg/min or 6mg/hr) will be infused during the ketamine periods, which is lower than required to induce sedation. No minimal sedation requirements will exist for the propofol or other regimen period. This will be done to test the effect of ketamine (which is hypothesized to affect frequency of SD) compared to other sedations regimens (which are not thought to affect SD.) Each period of adjustment of the sedation regimen will be treated as a "spontaneous breathing trial" which is a common standard of care procedure for nursing which involves holding sedation to determine a patient's neurologic exam and respiratory ability with subsequent titration back to appropriate clinical effect. These sedation breaks are very common in the ICU and titration to the desired clinical effect will be performed with the appropriate drug per the standard ICU nursing protocols. In the event that the patient no longer needs invasive positive pressure ventilation prior to discontinuation of ] neuromonitoring, propofol/other sedation intervals will not have mandatory sedative infusions, however, ketamine intervals will have a basal dose of 0.1mg/min (6mg/hr). 'The sedation protocol will end when the strip is removed. This is determined by the patients critical care needs. The strip is checked daily for function as well as any sign of problem such as leak of CSF. Once other critical care monitoring is discontinued (such as ventricular drains and invasive monitoring) the strip will be removed. Other endpoints will include any sign of CSF leak, adverse event reported, or treating intensivist does not think alternating sedation is safe.

During the sedation protocol, cortical electroencephalographic monitoring with the cortical electrodes will be continuously recording. Other physiologic data obtained clinically (including, but not limited to, vital signs, arterial wave forms, laboratory values, video EEG) will be subject to review and data collection for correlation with occurrence of SD. This data is obtained as part of standard of care and stored in a departmental server in an anonymous fashion. Clinical video EEG will be obtained on the majority of patients (if not all patients) as part of standard multimodal monitoring. This video will be reviewed to look for any external stimuli that might induce cortical spreading depressions.

ELIGIBILITY:
Inclusion Criteria:

* GCS <8
* SAH or severe traumatic brain injury requiring craniotomy
* Consent obtainable (via legal representative)
* Ictus (bleed or injury) within 48 hours of enrollment
* Clinically appropriate for multimodality monitoring

Exclusion Criteria:

* Anticipated survival <48 hours
* No craniotomy
* Infratentorial craniotomy only•Unable to obtain consent
* Absence of clinically used multimodality monitoring
* Prisoners
* Pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in frequency of Cortical Spreading depression with use of ketamine | approximately 7 days
  Frequency of events as defined by propagating slow potential change in adjacent leads with associated suppression of high frequency signal. Assessed by 2 experienced reviewers blinded to sedation arm.

SECONDARY OUTCOMES:
Change in frequency of Cortical Spreading depolarization with stimulation to patient | approximately 7 days
  Episodes of touching and other clinical manipulations will be scored by review of video EEG data and correlated with occurrence of CSD.
Change in frequency of Cortical Spreading depolarization with varying doses of ketamine | approximately 7 days
  CSD will be assessed as above, and if there is a response with Ketamine, a dose response assessment will be performed.
Presence of Scalp EEG tracings correlates to cortical spreading depolarization | approximately 7 days
  Using scalp EEG electrodes positioned above the cortical strip, propagating loss of high frequency signal in adjacent channels will be scored by an experienced EEG interpreter.
Correlation between pre-operative neurologic exam (GCS) and amount and frequency of cortical spreading depolarizations | approximately 7 days
  Glasgow Coma Scale score will be used.
Correlation between post-operative neurologic exam (GCS) and amount and frequency of cortical spreading depolarizations | approximately 7 days
  Glasgow Coma Scale will be used.
Subtype of CSD will be correlated with ketamine use. This includes Isoelectric, partially isoelectric, and clusters of CSD. | approximately 7 days
  Subtypes of CSD have previously been defined and will be scored by experienced reviewers using a standardized system. The outcome is "subtype of CSD" and so this single variable will be assessed for the effect of Ketamine.
Demographic factors associated with more frequent cortical depolarizations. | approximately 7 days
  Basic demographics including Age, Gender, injury type, and surgical procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Carlson, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Dreier JP, Isele T, Reiffurth C, Offenhauser N, Kirov SA, Dahlem MA, Herreras O. Is spreading depolarization characterized by an abrupt, massive release of gibbs free energy from the human brain cortex? Neuroscientist. 2013 Feb;19(1):25-42. doi: 10.1177/1073858412453340. Epub 2012 Jul 24. PMID 22829393
- [Background] Strong AJ, Fabricius M, Boutelle MG, Hibbins SJ, Hopwood SE, Jones R, Parkin MC, Lauritzen M. Spreading and synchronous depressions of cortical activity in acutely injured human brain. Stroke. 2002 Dec;33(12):2738-43. doi: 10.1161/01.str.0000043073.69602.09. PMID 12468763
- [Background] Fabricius M, Fuhr S, Bhatia R, Boutelle M, Hashemi P, Strong AJ, Lauritzen M. Cortical spreading depression and peri-infarct depolarization in acutely injured human cerebral cortex. Brain. 2006 Mar;129(Pt 3):778-90. doi: 10.1093/brain/awh716. Epub 2005 Dec 19. PMID 16364954
- [Background] Dohmen C, Sakowitz OW, Fabricius M, Bosche B, Reithmeier T, Ernestus RI, Brinker G, Dreier JP, Woitzik J, Strong AJ, Graf R; Co-Operative Study of Brain Injury Depolarisations (COSBID). Spreading depolarizations occur in human ischemic stroke with high incidence. Ann Neurol. 2008 Jun;63(6):720-8. doi: 10.1002/ana.21390. PMID 18496842
- [Background] Jeffcote T, Hinzman JM, Jewell SL, Learney RM, Pahl C, Tolias C, Walsh DC, Hocker S, Zakrzewska A, Fabricius ME, Strong AJ, Hartings JA, Boutelle MG. Detection of spreading depolarization with intraparenchymal electrodes in the injured human brain. Neurocrit Care. 2014 Feb;20(1):21-31. doi: 10.1007/s12028-013-9938-7. PMID 24343564
- [Background] Drenckhahn C, Winkler MK, Major S, Scheel M, Kang EJ, Pinczolits A, Grozea C, Hartings JA, Woitzik J, Dreier JP; COSBID study group. Correlates of spreading depolarization in human scalp electroencephalography. Brain. 2012 Mar;135(Pt 3):853-68. doi: 10.1093/brain/aws010. PMID 22366798
- [Background] Hartings JA, Wilson JA, Hinzman JM, Pollandt S, Dreier JP, DiNapoli V, Ficker DM, Shutter LA, Andaluz N. Spreading depression in continuous electroencephalography of brain trauma. Ann Neurol. 2014 Nov;76(5):681-94. doi: 10.1002/ana.24256. Epub 2014 Sep 17. PMID 25154587
- [Background] Nakamura H, Strong AJ, Dohmen C, Sakowitz OW, Vollmar S, Sue M, Kracht L, Hashemi P, Bhatia R, Yoshimine T, Dreier JP, Dunn AK, Graf R. Spreading depolarizations cycle around and enlarge focal ischaemic brain lesions. Brain. 2010 Jul;133(Pt 7):1994-2006. doi: 10.1093/brain/awq117. Epub 2010 May 26. PMID 20504874
- [Background] Dreier JP, Major S, Manning A, Woitzik J, Drenckhahn C, Steinbrink J, Tolias C, Oliveira-Ferreira AI, Fabricius M, Hartings JA, Vajkoczy P, Lauritzen M, Dirnagl U, Bohner G, Strong AJ; COSBID study group. Cortical spreading ischaemia is a novel process involved in ischaemic damage in patients with aneurysmal subarachnoid haemorrhage. Brain. 2009 Jul;132(Pt 7):1866-81. doi: 10.1093/brain/awp102. Epub 2009 May 6. PMID 19420089
- [Background] Hinzman JM, Andaluz N, Shutter LA, Okonkwo DO, Pahl C, Strong AJ, Dreier JP, Hartings JA. Inverse neurovascular coupling to cortical spreading depolarizations in severe brain trauma. Brain. 2014 Nov;137(Pt 11):2960-72. doi: 10.1093/brain/awu241. Epub 2014 Aug 24. PMID 25154387
- [Background] Bosche B, Graf R, Ernestus RI, Dohmen C, Reithmeier T, Brinker G, Strong AJ, Dreier JP, Woitzik J; Members of the Cooperative Study of Brain Injury Depolarizations (COSBID). Recurrent spreading depolarizations after subarachnoid hemorrhage decreases oxygen availability in human cerebral cortex. Ann Neurol. 2010 May;67(5):607-17. doi: 10.1002/ana.21943. PMID 20437558
- [Background] Feuerstein D, Manning A, Hashemi P, Bhatia R, Fabricius M, Tolias C, Pahl C, Ervine M, Strong AJ, Boutelle MG. Dynamic metabolic response to multiple spreading depolarizations in patients with acute brain injury: an online microdialysis study. J Cereb Blood Flow Metab. 2010 Jul;30(7):1343-55. doi: 10.1038/jcbfm.2010.17. Epub 2010 Feb 10. PMID 20145653
- [Background] Dreier JP, Woitzik J, Fabricius M, Bhatia R, Major S, Drenckhahn C, Lehmann TN, Sarrafzadeh A, Willumsen L, Hartings JA, Sakowitz OW, Seemann JH, Thieme A, Lauritzen M, Strong AJ. Delayed ischaemic neurological deficits after subarachnoid haemorrhage are associated with clusters of spreading depolarizations. Brain. 2006 Dec;129(Pt 12):3224-37. doi: 10.1093/brain/awl297. Epub 2006 Oct 25. PMID 17067993
- [Background] Hartings JA, Strong AJ, Fabricius M, Manning A, Bhatia R, Dreier JP, Mazzeo AT, Tortella FC, Bullock MR; Co-Operative Study of Brain Injury Depolarizations. Spreading depolarizations and late secondary insults after traumatic brain injury. J Neurotrauma. 2009 Nov;26(11):1857-66. doi: 10.1089/neu.2009.0961. PMID 19508156
- [Background] Hartings JA, Bullock MR, Okonkwo DO, Murray LS, Murray GD, Fabricius M, Maas AI, Woitzik J, Sakowitz O, Mathern B, Roozenbeek B, Lingsma H, Dreier JP, Puccio AM, Shutter LA, Pahl C, Strong AJ; Co-Operative Study on Brain Injury Depolarisations. Spreading depolarisations and outcome after traumatic brain injury: a prospective observational study. Lancet Neurol. 2011 Dec;10(12):1058-64. doi: 10.1016/S1474-4422(11)70243-5. Epub 2011 Nov 3. PMID 22056157
- [Background] Strong AJ, Hartings JA, Dreier JP. Cortical spreading depression: an adverse but treatable factor in intensive care? Curr Opin Crit Care. 2007 Apr;13(2):126-33. doi: 10.1097/MCC.0b013e32807faffb. PMID 17327732
- [Background] Sanchez-Porras R, Santos E, Scholl M, Stock C, Zheng Z, Schiebel P, Orakcioglu B, Unterberg AW, Sakowitz OW. The effect of ketamine on optical and electrical characteristics of spreading depolarizations in gyrencephalic swine cortex. Neuropharmacology. 2014 Sep;84:52-61. doi: 10.1016/j.neuropharm.2014.04.018. Epub 2014 May 4. PMID 24796257
- [Background] Sakowitz OW, Kiening KL, Krajewski KL, Sarrafzadeh AS, Fabricius M, Strong AJ, Unterberg AW, Dreier JP. Preliminary evidence that ketamine inhibits spreading depolarizations in acute human brain injury. Stroke. 2009 Aug;40(8):e519-22. doi: 10.1161/STROKEAHA.109.549303. Epub 2009 Jun 11. PMID 19520992
- [Background] Hertle DN, Dreier JP, Woitzik J, Hartings JA, Bullock R, Okonkwo DO, Shutter LA, Vidgeon S, Strong AJ, Kowoll C, Dohmen C, Diedler J, Veltkamp R, Bruckner T, Unterberg AW, Sakowitz OW; Cooperative Study of Brain Injury Depolarizations (COSBID). Effect of analgesics and sedatives on the occurrence of spreading depolarizations accompanying acute brain injury. Brain. 2012 Aug;135(Pt 8):2390-8. doi: 10.1093/brain/aws152. Epub 2012 Jun 19. PMID 22719001
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Background] Hocking G, Cousins MJ. Ketamine in chronic pain management: an evidence-based review. Anesth Analg. 2003 Dec;97(6):1730-1739. doi: 10.1213/01.ANE.0000086618.28845.9B. PMID 14633551
- [Background] Correll GE, Maleki J, Gracely EJ, Muir JJ, Harbut RE. Subanesthetic ketamine infusion therapy: a retrospective analysis of a novel therapeutic approach to complex regional pain syndrome. Pain Med. 2004 Sep;5(3):263-75. doi: 10.1111/j.1526-4637.2004.04043.x. PMID 15367304
- [Background] Elia N, Tramer MR. Ketamine and postoperative pain--a quantitative systematic review of randomised trials. Pain. 2005 Jan;113(1-2):61-70. doi: 10.1016/j.pain.2004.09.036. PMID 15621365
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Result] Carlson AP, Abbas M, Alunday RL, Qeadan F, Shuttleworth CW. Spreading depolarization in acute brain injury inhibited by ketamine: a prospective, randomized, multiple crossover trial. J Neurosurg. 2018 May 25;130(5):1513-1519. doi: 10.3171/2017.12.JNS171665. Print 2019 May 1. PMID 29799344